CLINICAL TRIAL: NCT01674894
Title: Kinetics in Time-lapse Culture of Human Preembryos
Brief Title: Study of the Cleavage of the Egg in Relation to the Stimulation Treatment
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000063
Record Dates: First submitted 2012-08-21; First posted 2012-08-29 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Female Infertility
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Women treated with Menopur
- Group 2: Women treated with Menopur and Bravelle

SUMMARY:
This post-marketing, single-center prospective study will be conducted in an open-label, non-interventional setting, for women seeking fertility treatment and will describe cleavage dynamics in relation to the age of the oocyte and gonadotrophin treatment.

ELIGIBILITY:
Inclusion Criteria:

1. IVF/ICSI treatment
2. Regular cycles of 25-35 days
3. Follicle stimulation with Bravelle and/or Menopur
4. Women aged 38-35 years
5. Long agonist or short antagonist treatment
6. Willing and able to understand a Danish, English or German patient information form
7. Willing and able to provide written Informed Consent

Exclusion Criteria:

1. BMI more than 35
2. Presence of hydrosalpinx on ultrasound
3. FSH more than 13 or antral follicle count (AFC) less than 4 at fertility investigation
4. Known allergic reactions to the planned medications
5. Use of testicular sperm

Ages: 38 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women suffering from infertility
Sampling Method: Non-Probability Sample
Enrollment: 356 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12-10 (Actual); Study Completion 2016-03-10 (Actual)

PRIMARY OUTCOMES:
Time to 2. polar body extrusion in transferred embryos (only Intracellular Sperm Injection) | Week 1 after oocyte retrieval
Time for disappearance of pronuclei in transferred embryos | Week 1 after oocyte retrieval
Time for first cleavage in transferred embryos | Week 1 after oocyte retrieval
Time for cleavage to 3-cell embryo and 4-cell embryo in transferred embryos | Week 1 after oocyte retrieval
Scoring of blastomere even-size, fragmentation and multinucleation at 4-cell stage | Week 1 after oocyte retrieval

SECONDARY OUTCOMES:
Total dose of gonadotrophin used | 1 month
Gonadotrophin dose per oocyte retrieved | 1 month
Number of oocytes retrieved | 1 month
Number of fertilized and cleaved oocytes | 1 month
Number of preembryos with top quality | 1 month
Implantation rate | 2 months
Ongoing pregnancy rate week 7 | 3 months
Live birth rate | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- Danish Fertility Clinic, Frederiksberg, Copenhagen, Denmark